CLINICAL TRIAL: NCT03011190
Title: Effectiveness of the Iconic Therapy in Youth With Suicidal Ideation/Self-injuring Behavior and Borderline Personality Traits: Study Protocol for a Randomized Controlled Trial
Brief Title: Effectiveness of the Iconic Therapy for Borderline Personality Disorder Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silvia Elisa Hurtado Santiago (Other)
Responsible Party: Sponsor-Investigator, Silvia Elisa Hurtado Santiago, Principal investigator, University of Malaga
Organization: University of Malaga (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: shs-ico-2015-01
Record Dates: First submitted 2016-12-28; First posted 2017-01-05 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Personality Disorder, Borderline
Keywords: Terapia Iconica; BPD; adolescence; suicide
MeSH Terms: conditions — Borderline Personality Disorder; Suicide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iconic Therapy (Experimental): The Iconic Therapy program consists of two parts: a) an intensive program of 10-12-week basic skills group 60-minute duration with a range of 6 to 8 face-to-face inserted sessions and b) an additional one-year program of 4 to 6 gradually less frequent face-to-face sessions. The groups are typically lead by two trainers -therapist and co-therapist- for about 8-12 outpatients. Added to these established sessions, a variable number of face-to-face individual sessions with the principal investigator will also take place. They will depend on participant´s requirements. They will consist on coaching their demands and providing human support throughout the study.
  Interventions: Behavioral: Emotional regulation
- Support therapy (Active Comparator): Support therapy consist of 10-12 weekly group sessions of 60-minute duration. Patients and trainers will learn and debate about different behavioral aspects of the borderline personality disorder: emotional instability and impulses control, Jacobson relaxation technique, self-image and communicational styles, mindfulness, self-esteem or social skills to name a few. The groups are typically lead by two trainers -therapist and co-therapist- for about 8-12 outpatients.Added to these established group sessions, a variable number of face-to-face individual sessions with the principal investigator will also take place. They will depend on participant´s requirements. They will consist on coaching their demands and providing human support throughout the study.
  Interventions: Behavioral: Emotional regulation

INTERVENTIONS:
Behavioral: Emotional regulation — Educate people with difficulty in regulating their emotions and help them acquire skills to do so

SUMMARY:
Borderline personality disorder (BPD) is the most prevalent personality disorder in young community population whose most severe complication is suicide. Pharmacotherapy should not be used as the primary treatment for BPD as the benefits are unclear. Psychotherapy is the main treatment for people with BPD and the current recommendation is adapting available comprehensive treatments to develop easier and briefer therapies that are also effective. Iconic Therapy is an innovative option whose good clinical results should be validated on a clinical trial.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) in the early adulthood is an increasing diagnosis among general population. First symptoms detection and early intervention might help prevent its aggravation and further BPD diagnosis. Iconic Therapy is an innovative manual-driven psychotherapy to specifically and intensively treat BPD symptoms. Preliminary clinical results are good. The aim of the present study is to assess the effectiveness of the Iconic Therapy in comparison to a support structured therapy in an ecological setting (Spanish public specialized mental health care). The study is planned as a randomized controlled prospective trial that will randomize 60 young people (15 to 25 years old) with suicidal ideation/self-injuring behaviour and borderline personality traits. Participants will be randomly assigned to one of the two groups: Iconic Therapy or support structured therapy on a 1:1 basis. Both the Iconic Therapy and the support therapy programs consist of 10-12 weekly sessions delivered by two trained psychologists for about 8-12 outpatients on group format. The primary outcome measure is the change of symptoms severity assessed by the Borderline Personality Disorder List (BSL-23). Secondary outcomes include suicidal ideation and behavior, non-suicidal self-injures maladjustment to the daily life and economic evaluation for health care. Assessments will be performed at baseline after the intervention 6 and 12 months of follow-up. It is hypothesized that those attending the Iconic Therapy group will show a permanently reduction of the severity of symptoms as compared with those attending the structured support group. Data will be analyzed using generalized estimating equations (GEE) models.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15-25 years old
* Suicidal ideation and/or self-injuring behavior
* BPD behavioural trends defined as the cut point for alarming BPD traits (>38 score) on Exploratory Questionnaire of Personality-III-BPD (CEPER-III-BPD)
* Sufficiently proficient in Spanish to follow the treatment

Exclusion Criteria:

* Antisocial personality disorder as measured in the Clinical Interview for Diagnostic and Statistical Manual (DSM-IV Axis II) (SCID-II)
* Substance or alcohol abuse
* High suicidal risk
* Negative expectations to be enrolled in the study as measured < 35 by the Expectation of Treatment Scale (ETS)

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change on the severity of borderline personality disorder measured by Borderline Personality Symptom List (BSL-23). | Baseline and up to 12 months after inclusion.
  This questionnaire (BSL-23) is a dimensional instrument: the most widely used to assess borderline personality disorder symptomatology improvement in clinical trials. The Spanish validated version of the questionnaire will be used.

SECONDARY OUTCOMES:
Sociodemographic variables | Baseline
  The following socio-demographic data will be collected: gender, age, marital status, parents´nationality, coexistence (no studies, primary studies, Secondary studies, University, Professional formation), occupation (student, working, both studying and working, pensioner) and family member or allied friend´s phone number for further contacts.
Change on the suicidal ideation and behavior measured by the Columbia Suicide History Form (SSRS). | Baseline and up to 12 months after inclusion.
  this instrument measures ideation (wish, thinking, intention and plan), ideation severity (frequency, duration, control capacity, disuasory elements and reasons) and suicidal behavior (attempts and acts). It is considered an adequate tool for treatment planning and research.
Change on non-suicidal self-injure diagnosis | Baseline and up to 12 months after inclusion.
  It does not exist a specific validated scale to assess non suicidal self injures so the investigators collected and asked about all the 6 Diagnostic and Statistical Manual (DSM-V) criteria. The investigators aim to separately describe the incidence of suicide attempts/acts vs non suicidal self injures in this study.
Change on the economic evaluation measured by the Client Service Receipt Inventory (CSRI) - adapted Spanish version (CSRI-Spanish version) | Baseline and up to 12 months after inclusion.
  Questionnaire to assess use of healthcare/social care services and other economic impacts. This instrument has two subscales to assess either direct costs (emergency services/hospital admissions use, specialised medical consultations, prescribed diagnosis trials and consumed medication) or indirect costs (absenteeism and quantity/quality of job performance on a 100-point scales).

OTHER OUTCOMES:
Change on the maladjustment to the daily life measured by the Maladjustment Scale (EI). | Baseline and up to 12 months after inclusion.
  It is a brief instrument of 6 self-report items assessing maladjustment to the daily life on psychiatric population. A six point Likert scale ranging from 0 (not at all) to 5 (very strong) is used. It is sensitive to therapeutic changes.
Satisfaction with the treatment assessed by the Opinion of treatment scale (OTS). | Through therapy completion, an average of 12 weeks.
  It is a quick and easy to administer 6-item scale for assessing satisfaction and rationale credibility : how believable, convincing and logical the treatment was from 0 (not at all) to 10 (very strong).
Change on the perceived subjective global improvement measured on a 7-point ad hoc Likert scale | Through therapy completion (an average of 12 weeks) and up to 12 months after inclusion
  Participants will be asked about their subjective impression : much/quite/little bit better, the same or much/quite/little bit worse compared to when they entered the study.
Change on family and friends´ perceived global improvement | Through therapy completion (an average of 12 weeks) and up to 12 months after inclusion
  Family and friend´s perceived global improvement will be asked on a 7-point ad hoc Likert scale: much/quite/little bit better, the same or much/quite/little bit worse compared to when they entered the study.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Bersabé, Psychologist, Study Chair — Malaga University; Fermín Mayoral, Psychiatrist, Study Director — Hospital Regional de Malaga
Locations (1):
- Silvia E. Hurtado-Santiago, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hurtado-Santiago S, Guzman-Parra J, Mayoral F, Bersabe RM. Iconic Therapy for the reduction of borderline personality disorder symptoms among suicidal youth: a preliminary study. BMC Psychiatry. 2022 Mar 29;22(1):224. doi: 10.1186/s12888-022-03862-x. PMID 35351048
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Hurtado-Santiago S, Guzman-Parra J, Bersabe RM, Mayoral F. Effectiveness of iconic therapy for the reduction of borderline personality disorder symptoms among suicidal youth: study protocol for a randomised controlled trial. BMC Psychiatry. 2018 Sep 3;18(1):277. doi: 10.1186/s12888-018-1857-x. PMID 30176878